CLINICAL TRIAL: NCT00994175
Title: A Randomized, Placebo-Controlled, Double-Blind Pilot Study of Pioglitazone Hydrochloride in Severe, Refractory Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 090244; 09-H-0244 (Other: The National Institutes of Health)
Record Dates: First submitted 2009-10-10; First posted 2009-10-14 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Severe, Refractory Asthma; Airway Inflammation; Airflow Obstruction
Keywords: Pioglitazone; Severe, Refractory Asthma; Peroxisome Proliferator-Activated Receptor Gamma; Airflow Obstruction; Airway Inflammation; Asthma
MeSH Terms: conditions — Asthma | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pioglitazone, Then Placebo (Experimental): Pioglitazone, 30 mg daily, was administered for the initial 2 weeks of the first treatment phase, followed by 45 mg daily for an additional 14 weeks. This was followed by a 4-week washout period. Subjects were assessed for clinical stability during a second 4-week run-in period prior to crossing over to the placebo phase for 16 weeks in the second treatment phase to receive the placebo.
  Interventions: Drug: Pioglitazone; Drug: Placebo
- Placebo, Then Pioglitazone (Experimental): Placebo was administered for 16 weeks. This was followed by a 4-week washout period. Subjects were assessed for clinical stability during a second 4-week run-in period prior to crossing over to the Pioglitazone treatment group. Pioglitazone, 30 mg daily, was administered for the initial 2 weeks of the treatment phase, followed by 45 mg daily for an additional 14 weeks.
  Interventions: Drug: Pioglitazone; Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone
Drug: Placebo

SUMMARY:
Background:

- Individuals who have severe asthma that is not easily controlled by current treatments are in need of new treatments to prevent potentially life-threatening asthma attacks. Experiments in mice have found that a medication called pioglitazone hydrochloride (Actos ), which is used to treat patients with diabetes, may be effective for treating severe asthma. Researchers are interested in determining whether Actos is effective in improving the quality of life in subjects with severe asthma who continue to have symptoms despite maximum standard medical therapy.

Objectives:

- To assess the effectiveness of pioglitazone hydrochloride as a treatment for patients with severe asthma that is not controlled by standard treatments.

Eligibility:

- Individuals between 18 and 75 years of age who have been diagnosed with and treated for severe asthma for at least 1 year.

Design:

* Potential participants will have a screening visit to determine eligibility for the study. The visit will involve breathing tests, chest x rays, heart and lung monitoring, and blood tests.
* Eligible participants will have a full medical history and will answer a series of questionnaires about their quality of life with asthma.
* Phase 1: Patients will record lung function and asthma symptoms morning and evening for 4 weeks. At the end of this period, patients will be evaluated with breathing, allergy, and blood tests, as well as questionnaires. Patients will also provide a sputum sample.
* Phase 2: Patients will receive regular doses of either pioglitazone hydrochloride or a placebo for 16 weeks. Patients will return to the National Institutes of Health every 4 weeks for tests.
* Phase 3: Wash-out period without study drugs for 4 weeks, similar to Phase 1.
* Phase 4: Patients will receive regular doses of either pioglitazone hydrochloride or a placebo for 16 weeks. Patients who received placebo will be given the study drug, and vice versa. Patients will return to the National Institutes of Health every 4 weeks for tests.
* Phase 5: Medications will be stopped, and patients will return to the National Institutes of Health 4 weeks later for final tests.

DETAILED DESCRIPTION:
New therapies are needed for patients with asthma who are sub-optimally controlled by standard measures. Pioglitazone hydrochloride (Actos ) is a highly selective and potent agonist for the peroxisome proliferator-activated receptor-Gamma (PPAR Gamma). Studies in murine models of allergic asthma have shown that PPAR Gamma agonists down-regulate allergen-mediated airway inflammation and airway hyperresponsiveness. This protocol is a randomized, placebo-controlled, doubleblind, crossover (phase II) pilot study of the efficacy of pioglitazone for the treatment of patients with severe, refractory asthma. The primary end-point for this study will be quality of life as determined by the Asthma Quality of Life Questionnaire (AQLQ) score. Secondary end-points will include indices of airway inflammation, airflow obstruction, airway hyperreactivity, and asthma symptoms.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects will be between 18 and 75 years of age, male or female, with a diagnosis of severe, refractory asthma, as defined by the American Thoracic Society, for at least one year.
* Subjects must have a history of reversible airflow obstruction as defined by a positive methacholine bronchoprovocation challenge or a positive response to inhaled bronchodilators at some point in the course of their disease or a greater than 20% variability in the Forced Expiratory Volume in 1 second (FEV1) or the peak expiratory flow (PEF) documented during serial measurements of lung function over time.
* Left ventricular ejection fraction greater than or equal to 50% by echocardiogram
* For women of childbearing potential, negative pregnancy test prior to study and willingness to adhere to reliable birth control methods during the study.
* Subjects must have the ability to provide informed consent

EXCLUSION CRITERIA:

* A known history of hypersensitivity to pioglitazone.
* Asthma exacerbation requiring treatment with additional oral corticosteroids in the previous 6 weeks, or a life-threatening asthma attack requiring cardiopulmonary support in the previous 6 months.
* Cigarette smoking within the previous 12 months or a prior history of > 20 cumulative pack-years.
* Investigational therapy for any indication within I month prior to the screening visit.
* History of lung disease other than asthma (ie., COPD, sarcoidosis).
* History of diabetes mellitus requiring treatment with any medication, insulin secreting tumor, or symptomatic hypoglycemia.
* HIV/AIDS
* History of congestive heart failure with current symptoms consistent with NYHA classification II, Ill or IV.
* Preexisting edema (2+ or greater).
* Hemoglobin < 11 gm/dl for males and < 10 gm/dl for females.
* Active liver disease or abnormal liver function tests > 2 times upper limit of normal.
* History of bladder or colon cancer.
* History of other cancer not in remission.
* Active breast feeding.
* Use of the following medications, which can interact with pioglitazone:

  * Gemfibrizol (Lopid)
  * Atazanivir (Reyataz)
  * Ritonavir (Norvir)
  * Rifampin (Rifadpin)
  * Carbamzepine (Tegretol)
  * Phenobarbital (Luminal)
  * Phenytoin (Dilantin)
  * Rifapentine (Priftin)
  * Secobarbital (Seconal)
  * Amiodarone (Cordarone, Pacerone)
  * Palitaxel (Taxol)
  * Replaglinide (Prandine)
  * Ketoconazole (Nizoral)
  * Atorvastatin (Lipitor )
  * Fosphenytoin (Cerebyx)
  * Itraconazole (Sporanox)
  * Trimethoprim (in Bactrim)
  * Thioridazine
* Certain over-the-counter herbs and supplements. These will be reviewed by the investigators for possible interactions with the study medication A determination of whether the supplement is safe to use with pioglitazone will be made on a case-by-case basis.
* Any condition that, in the investigator s opinion, places the patient at undue risk for complications from pioglitazone therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09-23; Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart J Levine, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - INOVA Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The NIH Biomedical Translational Research Information System

REFERENCES:
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Berry MA, Hargadon B, Shelley M, Parker D, Shaw DE, Green RH, Bradding P, Brightling CE, Wardlaw AJ, Pavord ID. Evidence of a role of tumor necrosis factor alpha in refractory asthma. N Engl J Med. 2006 Feb 16;354(7):697-708. doi: 10.1056/NEJMoa050580. PMID 16481637
- [Background] Erin EM, Leaker BR, Nicholson GC, Tan AJ, Green LM, Neighbour H, Zacharasiewicz AS, Turner J, Barnathan ES, Kon OM, Barnes PJ, Hansel TT. The effects of a monoclonal antibody directed against tumor necrosis factor-alpha in asthma. Am J Respir Crit Care Med. 2006 Oct 1;174(7):753-62. doi: 10.1164/rccm.200601-072OC. Epub 2006 Jul 13. PMID 16840747 (Retraction: PMID 21288870 Am J Respir Crit Care Med. 2011 Feb 1;183(3):418)
- [Result] Kaler M, Barochia AV, Weir NA, Cuento RA, Stylianou M, Roth MJ, Filie AC, Vaughey EC, Nathan SD, Levine SJ. A randomized, placebo-controlled, double-blinded, crossover trial of pioglitazone for severe asthma. J Allergy Clin Immunol. 2017 Dec;140(6):1716-1718. doi: 10.1016/j.jaci.2017.05.033. Epub 2017 Jun 15. PMID 28625806
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0244.html

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Started | 6 | 9
Completed | 4 | 8
Not Completed | 2 | 1
Period: Second Intervention
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Started | 4 | 8
Completed | 4 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All subjects who started the study.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 16 Weeks - Juniper Asthma Quality of Life Questionnaire (AQLQ) Score
Description: Juniper Asthma Quality of Life Questionnaire (AQLQ) score at the end of the pioglitazone treatment period as compared to the placebo treatment period. The AQLQ is scored on a 7-point scale with 7 = not impaired at all, 1 = severly impaired
Time Frame: 16 weeks
Population: All subjects who completed both treatment phases of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pioglitazone: Subjects received 30 mg daily of pioglitazone for the first 2 weeks of the treatment phase and then were escalated to 45 mg daily of pioglitazone for the 3rd through 16th weeks of the treatment phase
- Placebo: Subjects received a matched placebo.
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 4.7 (1.3) | 4.6 (1.3)

2. Primary Outcome: Baseline - Juniper Asthma Quality of Life Questionnaire (AQLQ) Score
Description: as for outcome 1
Time Frame: Baseline
Population: All subjects who completed both treatment phases of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 4.478 (0.9866) | 4.306 (1.342)

ADVERSE EVENTS:
Time Frame: 44 weeks
Arm/Group | Pioglitazone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 4/15
Other Adverse Events (participants affected / at risk) | 8/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=15) | Placebo (N=15)
Cataract (Eye disorders) | 0 | 1
Allergic oedema (General disorders) | 0 | 1
Allergic oedema (Immune system disorders) | 1 | 0
Oedema peripheral (Metabolism and nutrition disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=15) | Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Oral infection (Gastrointestinal disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Oedema (General disorders) | 3 | 1
Swelling (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Genitourinary symptom (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rabies immunisation (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes